CLINICAL TRIAL: NCT01547052
Title: Adapting Dialectical Behavior Therapy for Children in Residential Care: Pilot Randomized Clinical Trial With Children With Severe Emotional and Behavioral Dysregulation
Brief Title: Adapting Dialectical Behavior Therapy for Children in Residential Care
Acronym: DBT-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Green Chimneys Residential Treatment Center, Brewster, NY (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1012007764
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Childhood Aggression
Keywords: DBT, child, emotion regulation, behavior problems
MeSH Terms: conditions — Maple syrup urine disease, type 2; Emotional Regulation; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBT for children (Experimental): Dialectical Behavior Therapy adapted for children
  Interventions: Behavioral: DBT for children
- Enhanced Supportive-Educational Therapy (Active Comparator): Enhanced Treatment-As-Usual, including supportive-educational model, cognitive-behavioral skills and parent management training
  Interventions: Behavioral: Enhanced Supportive-Educational therapy

INTERVENTIONS:
Behavioral: DBT for children — intervention consists of weekly individual 45 min. sessions, twice per week 60 min. group sessions, and every other week 90 min. sessions with parents
  Other Names: Dialectical Behavior Therapy adapted for Children
  Arms: DBT for children
Behavioral: Enhanced Supportive-Educational therapy — weekly individual 45 min sessions, twice per week 60 min. group sessions and every other week parent sessions.
  Other Names: Enhansed TAU
  Arms: Enhanced Supportive-Educational Therapy

SUMMARY:
I: Conduct Pilot Randomized Clinical Trial of Dialectical Behavior Therapy for children (DBT-C) in residential as compared with Treatment-As-Usual (TAU) (60 children in DBT-C and 60 children in the comparison condition).

II: Finalize therapist training manuals and educational materials to guide selection, training, and supervision of treatment providers.

DETAILED DESCRIPTION:
Specific Aim 1: Examine feasibility of DBT-C by evaluating response rate in treatment attendance, treatment satisfaction, and any differences in these rates by groups.

Hypothesis 1: DBT-C will be equivalent to TAU in attendance rate and will have significantly greater treatment satisfaction rating by subjects, as well as by therapists and milieu staff.

Specific Aim 2: Examine efficacy of DBT-C as compared to TAU in reducing internalizing and externalizing symptoms.

Hypothesis 2: Children in DBT-C condition as compared to TAU will have significantly fewer internalizing and externalizing symptoms.

Specific Aim 3: Examine efficacy of DBT-C in improving adaptive coping, emotion regulation, risk taking, and social skills, and reducing depression.

Hypothesis 3: Children in DBT-C Training condition as compared to TAU will have significantly greater improvement in adaptive coping skills, emotion regulation, risk taking and impulsivity and social skills, and reducing depressive symptoms.

Specific Aim 4: Examine efficacy of DBT-C in reducing the frequency of critical incidents.

Hypothesis 4: Children in DBT-C condition as compared to TAU will have significantly fewer critical incidents, including psychiatric hospitalization, emergency room visits, total number of days inpatient, suicidal ideations and attempts, self-harm behaviors, sexual acting out, running away, stealing, police involvement, etc.

ELIGIBILITY:
Inclusion Criteria:

* age between 6 years 0 months and 12 years 11 months;
* male;
* in residential care at Green Chimneys;
* projected length of stay is at least 8 months.

Exclusion Criteria:

* pervasive developmental disorder;
* psychotic disorder;
* mental retardation; (all as per psychiatric evaluation at Green Chimneys);
* in care or custody of the Department of Social Services (DSS);
* caregivers do not speak English.

Ages: 6 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2011-04; Primary Completion 2015-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Attendance Form | post-treatment at 30 weeks

SECONDARY OUTCOMES:
Balloon Analog Risk Task | pre-treatment, week 6, 12, 18, 24, 30 of treatment and at 3 and 6 months follow-up
Mood and Feelings Questionnaire | pre-treatment, weeks 6, 12, 18, 24 and 30 of treatment at at 3 and 6 months follow-up
Emotion Regulation Checklist | pre-treatment, weeks 12, 24 and 30 of treatment at at 3 and 6 months follow-up
Children's Coping Strategies Checklist | pre-treatment, weeks 12, 24 and 30 of treatment at at 3 and 6 months follow-up
Pleasure Scale for Children | pre-treatment, weeks 12, 24 and 30 of treatment at at 3 and 6 months follow-up
Social Skills Rating Scale | pre-treatment, weeks 12, 24 and 30 of treatment at at 3 and 6 months follow-up
Therapy Satisfaction Questionnaire | week 30
Therapist Satisfaction Scale | week 30
Milieu Staff Satisfaction Questionnaire | every 6 months
Incident Report | pre-treatment, weeks 6, 12, 18, 24 and 30 of treatment at at 3 and 6 months follow-up
Psychosocial Treatment Compliance Scale | week 30
Child Behavior Checklist | at pre-treatment, 6, 12, 18, 24, 30 weeks of treatment, and at 3 and 6 months follow-up
Difficulty with Emotion Regulation Scale | pre-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Francheska Perepletchikova, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Green Chimneys Residential Treatment Center, Brewster, New York, United States